CLINICAL TRIAL: NCT04711967
Title: Prospective Study of Fecal Microbiota Transplantation for Acute Intestinal GVHD After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Prospective Study of FMT for Acute Intestinal GVHD After Allo-HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020SDUCRCC015
Record Dates: First submitted 2020-12-30; First posted 2021-01-15 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-01

CONDITIONS: Acute Graft Versus Host Disease in Intestine
Keywords: Acute-graft-versus-host Disease; Fecal microbiota transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation group (Experimental): treat with FMT
  Interventions: Biological: Fecal Microbiota Transplantation
- Control group (Active Comparator): treat with traditional medicine
  Interventions: Drug: drug

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — fecal microbiota transplantation
  Arms: Fecal Microbiota Transplantation group
Drug: drug — drug
  Arms: Control group

SUMMARY:
Acute intestinal GVHD is the main cause of death after allo-HSCT, and FMT is a new treatment method for this disease. In this prospective study, the investigators will recruit intestinal GVHD patients to demonstrate the efficacy and safety of FMT.

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) is a common complication of allogeneic hematopoietic stem cell transplantation (allo-HSCT), of which intestinal GVHD is a particularly serious one, which is the main cause of death after allo-HSCT. Recent studies have demonstrated that intestinal flora imbalance is strongly associated with the risk of infection and mortality in patients with allo-HSCT. On the basis of this theory, fecal microbiota transplantation (FMT) may be an effective method for GVHD, that is, fecal suspension from healthy individuals is inputted into the digestive tract of patients through some methods, so as to restore the microbial community diversity of patients. In this prospective study, the investigators aimed to demonstrate the efficacy and safety of this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. received allo-HSCT due to a hematopoietic disease
2. corticosteroid resistant/dependent intestinal GVHD
3. ECOG≤2
4. Sign informed Consent
5. No major organ dysfunction

Exclusion Criteria:

1. uncontrolled or severe infections
2. patients with severe liver and kidney function, cardiopulmonary insufficiency, epilepsy, and central nervous system disorder
3. high-risk bleeding
4. ANC<0.5×10^9/L or PLT<20x10^9/L
5. hepatitis B, tuberculosis, syphilis, and HIV antibody positive or acute phase of any infectious disease
6. patients participating in other clinical trials
7. patienta who suffer from mental illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change in times of stool | day 0,day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 14, day 21 and day 28.
  Change in times of stool per day within 28 days after FMT
change in volume of stool | day 0,day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 14, day 21 and day 28.
  Change in volume of stool per day within 28 days after FMT

SECONDARY OUTCOMES:
Change in life quality up to 28 days | day 0,day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 14, day 21 and day 28.
  The change quality of patients life within 28 days after FMT is assessed by "EORTC Quality of Life measurement Scale QLQ-C30 (V3.0)" with a score ranged 0~100. And the higher the score, the better the functional status and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Shuqian Xu, Principal Investigator — Qilu Hospital of Shandong University
Locations (2):
- China (2):
  - Peking university people's hospital, Beijing, Beijing Municipality
  - Shandong university qilu hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No